CLINICAL TRIAL: NCT00268606
Title: Tailored Cognitive-Behavioral Therapy for Fibromyalgia Patients at Risk: A Randomized, Controlled Trial
Brief Title: Tailored Cognitive-Behavioral Therapy for Fibromyalgia Patients at Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Collaborators: Reumafonds (Unknown); Radboud University Medical Center (Other); Sint Maartenskliniek (Other)
Organization: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60-00636-98-028; NR 05-1-1101
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; cognitive-behavioral therapy; tailored treatment
MeSH Terms: conditions — Fibromyalgia | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: cognitive-behavioral therapy

SUMMARY:
The present study is a new approach of examining tailored cognitive-behavioral interventions for fibromyalgia patients at risk. For this purpose, fibromyalgia patients are screened with respect to cognitive-behavioral risk factors and these patients are offered tailored cognitive-behavioral treatment options. It is expected that this approach will result in increased magnitude and maintenance of effects.

DETAILED DESCRIPTION:
The fibromyalgia syndrome is a chronic condition with widespread pain that poses a great challenge for patients, rheumatologists and society because of the lack of optimal treatment options. There is extensive evidence that, in comparison with patients with rheumatoid arthritis, fibromyalgia patients report higher levels of functional disability, pain, fatigue, and lower levels of quality of life. Although effectiveness of pharmacological agents and other interventions is generally limited, most promising effects have been found for non-pharmacological treatments, particularly those with a primary focus on cognitive-behavioral treatment components. However, also these treatment outcomes are characterized by large individual variation. Particularly patients with less impairments in daily life seem to benefit less from these treatments. In line with the international literature, previous findings of the research group suggest that effectiveness might be increased when tailored cognitive-behavioural treatments are solely offered to patients at risk.

In the present project the effects of tailored interventions based on cognitive-behavioral factors for patients at risk are studied. In a randomized, controlled trial, fibromyalgia patients are screened for risk profiles. Patients at risk will be assigned to tailored cognitive or behavioral treatment conditions, depending on their risk profile with respect to cognitive-behavioral factors. Half of the patients are subsequently randomly assigned to a waiting list control condition. It is expected that this tailored treatment approach will increase magnitude and maintenance of treatment effects for pain, disability, fatigue and increased quality of life, which means an important step forward for patients, involved professionals and society.

ELIGIBILITY:
Inclusion Criteria:

* fibromyalgia according to the criteria of the American College of Rheumatology (ACR)

Exclusion Criteria:

* physical or psychological comorbidity that interferes with cognitive-behavioral treatment
* participation in other clinical trials
* other psychological treatments
* pregnancy
* illiteracy
* difficulties with understanding Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2003-12; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
pain
disability
fatigue
psychological distress at post treatment and 6 month follow-up

SECONDARY OUTCOMES:
passive coping
illness cognitions
social support at post treatment and 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: A.W.M. Evers, Phd, Study Chair — Radboud University Nijmegen Medical Centre, department of Medical Psychology; F.W. Kraaimaat, Prof. Phd, Study Chair — Radboud University Nijmegen Medical Centre, deparment of Medical Psychology; W. van Lankveld, Phd, Study Chair — Sint Maartenskliniek, department of Reseach and Development
Locations (5):
- Netherlands (5):
  - Jeroen Bosch Ziekenhuis, department of Medical Psychology, 's-Hertogenbosch
  - Rijnstate Hospital, department of Rheumatology, Arnhem
  - Radboud University Medical Centre, department of Rheumatology, Nijmegen
  - Radboud University Nijmegen Medical Centre, department of Medical Psychology, Nijmegen
  - Sint Maartenskliniek, Nijmegen

REFERENCES:
- [Derived] van Koulil S, van Lankveld W, Kraaimaat FW, van Helmond T, Vedder A, van Hoorn H, Donders AR, Wirken L, Cats H, van Riel PL, Evers AW. Tailored cognitive-behavioural therapy and exercise training improves the physical fitness of patients with fibromyalgia. Ann Rheum Dis. 2011 Dec;70(12):2131-3. doi: 10.1136/ard.2010.148577. Epub 2011 Sep 16. PMID 21926189
- [Derived] van Koulil S, Kraaimaat FW, van Lankveld W, van Helmond T, Vedder A, van Hoorn H, Donders AR, Thieme K, Cats H, van Riel PL, Evers AW. Cognitive-behavioral mechanisms in a pain-avoidance and a pain-persistence treatment for high-risk fibromyalgia patients. Arthritis Care Res (Hoboken). 2011 Jun;63(6):800-7. doi: 10.1002/acr.20445. PMID 21312345
- [Derived] van Koulil S, van Lankveld W, Kraaimaat FW, van Helmond T, Vedder A, van Hoorn H, Donders R, de Jong AJ, Haverman JF, Korff KJ, van Riel PL, Cats HA, Evers AW. Tailored cognitive-behavioral therapy and exercise training for high-risk patients with fibromyalgia. Arthritis Care Res (Hoboken). 2010 Oct;62(10):1377-85. doi: 10.1002/acr.20268. PMID 20521308
- [Derived] van Koulil S, Kraaimaat FW, van Lankveld W, van Riel PL, Evers AW. A patient's perspective on multidisciplinary treatment gain for fibromyalgia: an indicator for pre-post treatment effects? Arthritis Rheum. 2009 Dec 15;61(12):1626-32. doi: 10.1002/art.24792. PMID 19950305